CLINICAL TRIAL: NCT03572816
Title: The Effect of a Heel-unloading Orthosis in Short-term Treatment of Calcaneus Fractures on Physical Function, Quality of Life and Return to Work - a Randomized Controlled Trial
Brief Title: Heel-unloading Orthosis for Treatment of Calcaneus Fractures
Acronym: CALCFRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20170219
Record Dates: First submitted 2018-05-28; First posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Calcaneus Fracture; Orthopedic Devices Associated With Misadventures

STUDY DESIGN:
Intervention Model Description: The study design is a parallel group, randomized controlled trial with open allocation including all patients with calcaneus fractures independent of kind of initial therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current standard (No Intervention): * mobilization without weight bearing for 6 weeks starting with the day of either decision-making for non-operative therapy or open reduction and internal fixation, if needed a cast or another kind of orthosis as a Static Walker are applied, then 4 weeks 15-20 kg, 2 weeks 35-45 kg, after that transition to full-weight bearing (always only if possible)
  * X-ray after 6 and 12 weeks; depending on the results, the schedule for weight bearing may be adjusted to the need in case of delayed healing or complications related to implants
- Intervention (Experimental): * mobilization with the custom-made heel-unloading orthosis ('Settner shoe') without pads for 6 weeks, then 2 weeks one pad, 2 weeks 2 pads, 2 weeks 3 pads, after that full-weight bearing without any support (always only if possible)
  * X-ray after 6 and 12 weeks; depending on the results, the schedule for weight bearing may be adjusted to the need in case of delayed healing or complications related to implants
  Interventions: Device: Settner shoe

INTERVENTIONS:
Device: Settner shoe — custom-made heel-unloading orthosis ('Settner shoe') in aftercare of calcaneus fractures (used according to manufacturer), certified 'CE' product with more than 10 years experience
  Arms: Intervention

SUMMARY:
Treatment of acute calcaneus fractures includes non- or partial weight bearing, but protocols are different and often not very specific. In fact, there are no studies published comparing different procedures or special supporting devices. Recently, a heel-unloading orthosis ('Settner shoe') was introduced, allowing walking by shifting the load to the middle- and forefoot. Specifically in calcaneus fractures, early regain of physical activity has been highlighted as one of the key factors for quality of life and the ability to return to work. Thus, the investigators hypothesize that mobilization with the 'Settner shoe' results in higher physical activity within the first 3 months and secondly improves ability to return to work in calcaneus fracture patients aged 18-60 years.

DETAILED DESCRIPTION:
In the past decades, the scientific focus regarding calcaneus fractures was the choice of operative or non-operative treatment modality. Although the evidence is ambiguous, recent meta-analyses suggest that operative therapy is associated with a higher likelihood to resume pre-injury work, to reach a higher level of physical function and fewer problems when wearing shoes. However, non-operative therapy has significant less complications and infections. Typically, aftercare includes non- or partial weight bearing, but protocols are different and often not very specific. In fact, there are no studies published comparing different procedures or special supporting devices. Recently, a heel-unloading orthosis ('Settner shoe') was introduced in aftercare for calcaneus fractures, allowing walking by shifting the load to the middle- and forefoot. This orthosis does not only enable early mobilization of patients suffering one-sided fractures, but also permits going following two-sided fractures, avoiding the otherwise necessary wheel-chair mobilization. The 'Settner shoe' can be applied in non-operative therapy and following operations. Specifically in calcaneus fractures, early regain of physical activity has been highlighted as one of the key factors for quality of life and the ability to return to work. Thus, the investigators hypothesize that mobilization with the 'Settner shoe' results in higher physical activity within the first 3 months and secondly improves ability to return to work in calcaneus fracture patients aged 18-60 years. Further outcome criteria are the American Orthopaedic Foot and Ankle Society's (AOFAS) ankle-hindfoot assessment, a 3-dimensional gait analysis, and the EQ-5D-3L questionnaire. It is the first trail applying a standardized aftercare in patients suffering from calcaneus fractures aiming to improve the non-operative part of treatment. Furthermore, the trial clarifies, whether the economical effort for the equipment acquisition is scientifically justified.

The investigators hypothesize that mobilization with the 'Settner shoe' results in higher physical activity within the first 3 months after calcaneus fractures.

Research questions

Does the application of a heel-unloading orthosis ('Settner shoe') independent of operative or non-operative therapy of a calcaneus fracture improve:

1. the physical activity (active minutes per day)?
2. the quality of life (EQ-5D-3L)?
3. the foot function (AOFAS)?
4. the time necessary for return to work in patients between 18 and 60 years?

ELIGIBILITY:
Inclusion Criteria:

* Fracture of the calcaneus, which is classifiable according to the Sanders' classification (excludes avulsion fractures)
* Being able to understand Danish or English and answer the questionnaires
* Informed consent

Exclusion Criteria:

* Pathological fractures
* Immature skeletal system
* Other fractures with influence on weight-bearing
* A soft-tissue situation not allowing the equipment with a 'Settner shoe' within 3 weeks after treatment (either decision-making for non-operative therapy or open reduction and internal fixation)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
activity | 3 months
  the number of active minutes per day

SECONDARY OUTCOMES:
QoL | 3 months
  the EuroQol 5D-3L questionnaire following
QoL | 6 months
  the EuroQol 5D-3L questionnaire following
activity | 6 months
  the number of active minutes per day

OTHER OUTCOMES:
AOFAS | 3 months
  functional foot score, The American Orthopedic Foot and Ankle Score, includes pain, function, alignment, for AOFAS calculation the subscores are added, ranges between 0 (worst) and 100 (best) points
AOFAS | 6 months
  functional foot score, The American Orthopedic Foot and Ankle Score, includes pain, function, alignment, for AOFAS calculation the subscores are added, ranges between 0 (worst) and 100 (best) points
Gait | 3 months
  3-dimensional gait analysis
Work | 6 months
  time point of return to work
Range of motion (ROM) | 3 months
  Pro- and supination (percent of healthy side or assumed normal mobility) are analyzed.
Range of motion (ROM) | 6 months
  Pro- and supination (percent of healthy side or assumed normal mobility) are analyzed.
pain | 3 months
  The subjective pain of patients is assessed using a Visual Analog Scale (VAS) in combination with registration of their pain medication, which is classified according to the WHO pain ladder. The Summary Pain Score (SPS) is calculated from the sum of the two components.
  VAS 0 (best) - 10 (worst) WHO scale for pain medication 0 (best, lowest) - 5 (worst, highest)
pain | 6 months
  The subjective pain of patients is assessed using a Visual Analog Scale (VAS) in combination with registration of their pain medication, which is classified according to the WHO pain ladder. The Summary Pain Score (SPS) is calculated from the sum of the two components.
  VAS 0 (best) - 10 (worst) WHO scale for pain medication 0 (best, lowest) - 5 (worst, highest)

CONTACTS AND LOCATIONS:
Overall Officials: Hagen Schmal, Prof, Principal Investigator — University Hospital Odense, Department of Orthopaedic Surgery
Locations (1):
- University Hospital Odense, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan, may come.

REFERENCES:
- [Background] Bruce J, Sutherland A. Surgical versus conservative interventions for displaced intra-articular calcaneal fractures. Cochrane Database Syst Rev. 2013 Jan 31;(1):CD008628. doi: 10.1002/14651858.CD008628.pub2. PMID 23440830
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Sanders R. Intra-articular fractures of the calcaneus: present state of the art. J Orthop Trauma. 1992;6(2):252-65. doi: 10.1097/00005131-199206000-00022. No abstract available. PMID 1602349
- [Derived] Schmal H, Larsen AH, Froberg L, Erichsen JL, Madsen CF, Pedersen L. The effect of a heel-unloading orthosis in short-term treatment of calcaneus fractures on physical function, quality of life and return to work - study protocol for a randomized controlled trial. Trials. 2019 Jun 4;20(1):324. doi: 10.1186/s13063-019-3447-8. PMID 31164153

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT03572816/Prot_SAP_000.pdf
  • Informed Consent Form: original version in Danish (2017-12-26): https://cdn.clinicaltrials.gov/large-docs/16/NCT03572816/ICF_001.pdf
  • Informed Consent Form: translated version in English (2017-12-26): https://cdn.clinicaltrials.gov/large-docs/16/NCT03572816/ICF_002.pdf